CLINICAL TRIAL: NCT02863094
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment for Schizophrenia Patients With Auditory Hallucinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSFC-81171273-01
Record Dates: First submitted 2016-07-07; First posted 2016-08-11 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Schizophrenia; Transcranial Magnetic Stimulation; Functional Magnetic Resonance Imaging
Keywords: schizophrenia; auditory hallucinations; functional magnetic resonance imaging; transcranial magnetic stimulation
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Stimulation (Active Comparator): The continuous theta burst stimulation (cTBS) protocol lasted 40 s and consisted of burst of 3 pulses delivered at 50 Hz, with bursts being repeated every 200 ms (at 5 Hz) for a total of 600 pulses. In the cTBS session, this 40s protocol was repeated for three times (1800 pulses in total) separated by two 15 min breaks (controlled by a stopwatch). MRI dataset should be acquired before the first cTBS session and after the last cTBS session.
  Interventions: Device: transcranial magnetic stimulation
- Placebo Stimulation (Sham Comparator): The procedure of this protocol was performed by a placebo coil. Each session lasted 40 s and consisted of burst of 3 pulses delivered at 50 Hz, with bursts being repeated every 200 ms (at 5 Hz) for a total of 600 pulses. No actual magnetic stimulation was applied on the head of the volunteers. MRI dataset should be acquired before the first sham TBS session and after the last sham TBS session.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation

SUMMARY:
To investigate the treatment effect of continuous transcranial magnetic stimulation on schizophrenia patients with auditory hallucinations, and the underlying neural mechanism by functional MRI

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after repetitive transcranial magnetic stimulation (rTMS) treatment. Patients were randomly allocated to rTMS group and the sham group by random number. There are about 30 patients in each group.The decision to enroll a patient was always made prior to randomization. Patients were studied using a double-blind design. Study participants, clinical raters, and all personnel responsible for the clinical care of the patient remained masked to allocated condition and allocation parameters. Only rTMS administrators had access to the randomization list; they had minimal contact with the patients, and no role in assessing AVH and other measures. Each patient would be treated for continuous 15 days by rTMS

Before the rTMS treatment, the Auditory Hallucination Rating Scale, Psychotic Symptom Rating Scale, and the Positive and Negative Syndrome Scale were obtained by a trained investigator to assess baseline severity of auditory verbal hallucination (AVH) and other symptoms. The patients had receiving a battery measure of neuropsychological tests (standardized tests to investigate their cognitive problems, anxiety and depressive symptoms in daily life), magnetic resonance imaging scan in multimodalities, electroencephalography (EEG), event-related potentials during stop signal test and Iowa-gambling test record.

After the last treatment, the Auditory Hallucination Rating Scale, Psychotic Symptom Rating Scale, and the Positive and Negative Syndrome Scale were obtained, as well as the Global Index of Safety to assess adverse events of the treatment. Patients were instructed to focus their answers on the past 15 days. The patients had also receiving a battery measure of neuropsychological tests, magnetic resonance imaging scan in multimodalities, and EEG record.

A month after the last treatment, participants were interviewed to obtain the Auditory Hallucination Rating Scale, Psychotic Symptom Rating Scale, the Positive, and Negative Syndrome Scale. They were instructed to focus their answers on the past week. Additionally, they were also asked to assess the battery of neuropsychological tests, and have magnetic resonance imaging scan in multimodalities, and EEG record. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Patients met diagnostic criteria for schizophrenia or schizoaffective disorder using the Structural Clinical Interview for Diagnostic and Statistical Manual Diploma in Social Medicine (DSM)-IV (SCID, Version 2.0),
* Patients reported auditory hallucinations at least 5 times per day based on pre-enrollment assessments using a written log or hand-held counter.
* Patients remain their psychotropic medication at steady dosages for at least 4 weeks prior to study entry and for the duration of the trial.
* Verbal intelligence quotient > 85 as measured by using a Chinese version of the National Adult Reading Test.

Exclusion Criteria:

* History of significant head trauma or neurological disorders
* Alcohol or drug abuse
* Focal brain lesions on T1- or T2-weighted fluid-attenuated inversion-recovery magnetic resonance images
* a prior history of a seizure not induced by drug withdrawal,
* first degree relative with epilepsy, significant neurological illness or head trauma, endocrine disease, such as thyroid disease, significant unstable medical condition,
* recent aggression or other forms of behavioral dyscontrol
* left-handedness, pregnancy
* estimated intelligence quotient<80
* current alcohol or drug abuse
* inability to provide informed consent.
* Hamilton Anxiety Rating Scale or the Hamilton Depression Rating Scale score > 7

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Symptom improvement assessed by Auditory Hallucination Rating Scale | up to 2 months

SECONDARY OUTCOMES:
functional connectivity of the temporal parietal junction assessed by functional MRI | up to 2 months
  Functional MRI measures: the functional connectivity between stimulated target and the whole brain areas
Global network properties assessed through Graph Theory | up to 2 months
Symptom improvement assessed by Positive and Negative Syndrome Scale | up to 2 months
Global structural connectivity assessed by diffusion weighted image | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, MD, Principal Investigator — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hua Q, Wang L, He K, Sun J, Xu W, Zhang L, Tian Y, Wang K, Ji GJ. Repetitive Transcranial Magnetic Stimulation for Auditory Verbal Hallucinations in Schizophrenia: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2444215. doi: 10.1001/jamanetworkopen.2024.44215. PMID 39527055